CLINICAL TRIAL: NCT07034989
Title: Investigation of the Effectiveness of Telerehabilitation-Assisted Exercise Training in Individuals With Rheumatoid Arthritis-Associated Interstitial Lung Disease
Brief Title: Effectiveness of Telerehabilitation-Assisted Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zülal TATAR (Other)
Responsible Party: Sponsor-Investigator, Zülal TATAR, Researcher, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Telerehabilitation ILD-RA
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Telerehabilitation; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asynchronous exercise group (Active Comparator)
  Interventions: Other: Exercise
- Control Group (No Intervention)

INTERVENTIONS:
Other: Exercise — Teach respiratory exercises and function-focused trunk stabilization exercises to individuals with RA-IAH via online platforms. Subsequently, instructional exercise videos will be delivered to the patients online. The respiratory exercise training will include thoracic expansion and diaphragmatic breathing exercises. The program will consist of a warm-up phase including 10 minutes of trunk stabilization exercises, a 40-minute functional exercise session targeting the upper and lower extremities with trunk stabilization, followed by a cooldown phase including 10 minutes of flexibility exercises involving trunk stabilization. The exercise videos related to these phases will be sent to the participants online. Participants will start the exercises with 6 repetitions and will be encouraged to increase to 8 repetitions as the program progresses. The assigned physiotherapist will contact patients once a week by phone to monitor exercise adherence.
  Arms: Asynchronous exercise group

SUMMARY:
This study aimed to evaluate the effectiveness of asynchronously implemented telerehabilitation-supported respiratory physiotherapy and function-oriented trunk stabilization exercises, which have not been previously applied in individuals with RA-IAH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA according to the 2010 EULAR/American College of Rheumatology diagnostic criteria
* Individuals with RA-associated Interstitial Lung Disease
* Individuals aged ≥18
* Agreeing to attend regular training throughout the study
* Having access to the internet and a computer

Exclusion Criteria:

* 10 pack-year smoking history
* Surgery or arthroscopic surgery within the last year
* Having any neurological or psychological disease that may prevent participation
* Patient's inability to comply with evaluation and education
* Having a psychiatric disease that will affect cooperation
* Individuals with serious functional limitations and cardiopulmonary and/or neurological disease unrelated to RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation Measurement | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.

SECONDARY OUTCOMES:
Evaluation of respiratory muscle strength | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
Modified Borg Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  Although it is frequently used today to define the severity of exertional dyspnea, it is also a scale that can be used to evaluate the severity of resting dyspnea. It consists of ten items that define the severity of dyspnea according to their degrees.
Modified Medical Research Council Dyspnea Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  It is a scale based on various physical activities that cause dyspnea. It consists of five items. The patient rates respiratory distress between 0 (no shortness of breath) and 4 (shortness of breath during activities such as being homebound and dressing).
Visual Analog Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  It consists of a 100 mm long horizontal line with the words "none" and "very severe" written on one end. The patient marks the severity of the current respiratory distress on the line using these two degrees as criteria. Scoring is done by measuring the marked area with the help of a tape measure.
Leicester Cough Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  Measures the effect of cough on quality of life. It consists of 19 questions. It has psychological, social and physical sub-dimensions. The cut-off value of the scale is not defined; low scores indicate being more affected by cough, i.e. worse quality of life.
St. George's Respiratory Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  It will be used to evaluate the health-related quality of life of the cases. SGRQ consists of three categories where the symptoms, activities and the effects of the disease on their daily lives are evaluated. The symptoms examined are cough, sputum, wheezing and shortness of breath. Physical functions, housework and hobbies are questioned to determine the activity status. These are activities limited by shortness of breath. The survey consisting of a total of 76 questions is completed in 20 minutes. There is an evaluation scale between zero and 100 points. Zero indicates perfect health status, 100 indicates the worst health status.
Short Form-36 Quality of Life Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  Short form-36 is a quality of life scale consisting of 36 items that can be filled by the patient and whose validity and reliability have been shown in studies in patients with musculoskeletal disorders. The Turkish version of SF-36 was used in our study. This scale includes 8 separate health-related headings as physical function (10 items), social function (2 items), physical role limitation (4 items), emotional role limitation (3 items), mental health (5 items), vitality (4 items), pain (2 items), general health (6 items).
Health Assessment Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  Since it evaluates activities of daily living comprehensively and in all dimensions, HAQ was preferred in our study to assess the disability level. It includes 20 questions across 8 domains (dressing, arising, eating, walking, hygiene, reach, grip, and common activities). Each question is scored between 0 and 3 (without any difficulty = 0, with some difficulty = 1, with much difficulty = 2, unable to do = 3). The highest score of each subsection is summed up and divided by 8 to determine the total score between 0 and 3. A high score indicates a low functional level
Disease Activity | Evaluations started immediately after receiving ethics committee approval and will be completed within 3 months, which is the study period.
  Disease activity in rheumatoid arthritis will be assessed using the Clinical Disease Activity Index (CDAI). This index is calculated based on four main parameters: the number of painful joints, the number of swollen joints, the visual analog scale of global disease activity as assessed by the patient, and the visual analog scale of global disease activity as assessed by the physician. CDAI scores of 0-2.8 indicate remission, 2.9-10 indicate low disease activity, 11-22 indicate moderate activity, and 22-76 indicate high activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Malatya, Turkey (Türkiye)